CLINICAL TRIAL: NCT06642363
Title: The Effectiveness of Astaxanthin Supplementation on the Clinical Symptoms and Cardio-metabolic Profile in Women with Polycystic Ovary Syndrome: a Protocol for a Randomized Double-blinded, Placebo-controlled Parallel-group Study
Brief Title: The Effectiveness of Astaxanthin Supplementation on the Clinical Symptoms and Cardio-metabolic Profile in Women with Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Milad Nasiri Jounaghani, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: IR.MUI.RESEARCH.REC.1402.204
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: PCO - Polycystic Ovaries; Obesity and Obesity-related Medical Conditions
Keywords: Astaxanthin; Polycystic Ovary Syndrome; Obesity; Hirsutism
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Hirsutism

STUDY DESIGN:
Intervention Model Description: Masking In this study, the individual conducting the blood test, the one prescribing the supplements, and the person analyzing the data are unaware of the division of participants into two groups: drug and placebo. Since the astaxanthin supplement and placebo are identical in color and shape, patients are also unaware of this division.
  Blinding All baseline assessments will be conducted before randomization, and certain assessments will be performed with blinding for group allocation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In this study, the individual conducting the blood test, the one prescribing the supplements, and the person analyzing the data are unaware of the division of participants into two groups: drug and placebo. Since the astaxanthin supplement and placebo are identical in color and shape, patients are also unaware of this division.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug (Experimental): receiving ASX supplements
  Interventions: Drug: Subjects in the intervention group will receive one capsule containing 10 mg Astaper day made by the "Zyest Technology Tarawat Zendig" institute in Iran. The dosage of ASX is determined based on the s
- control (Placebo Comparator): receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Subjects in the intervention group will receive one capsule containing 10 mg Astaper day made by the "Zyest Technology Tarawat Zendig" institute in Iran. The dosage of ASX is determined based on the s — Subjects in the intervention group will receive one capsule containing 10 mg Astaper day made by the "Zyest Technology Tarawat Zendig" institute in Iran. The dosage of ASX is determined based on the s
  Arms: Drug
Drug: Placebo — The placebo group will take one capsule containing corn starch in a wrapped and covered form and the appearance of ASX supplementation (blinding).
  Arms: control

SUMMARY:
Abstract Background: This trial aims to investigate the effect of 12 weeks of 10 mg/day astaxanthin (ASX) administration compared with the control group on insulin sensitivity, lipid profile, circulating MDA levels, severity of hirsutism, and depression in women with Polycystic Ovary Syndrome (PCOS).

Methods: This manuscript will outline the design, methodology, and potential clinical implications of ASX supplementation in eligible women with PCOS and a body mass index of 25-35 kg/m2, who are referred to the gynecologist clinic in Isfahan, Iran, during 2024-2025.

Discussion: This study is one of the first attempts to assess the clinical efficacy of astaxanthin as an auxiliary treatment in PCOS patients, and will provide more evidence in this area.

Trial registration number: Iran Clinical Trials (IRCT) website. (IRCT20231001059573N1)

DETAILED DESCRIPTION:
Introduction Polycystic Ovary Syndrome (PCOS) is a significant endocrine disorder affecting women of reproductive age, associated with common symptoms, including anovulation, infertility, metabolic dysfunction, cardiovascular issues, dyslipidemia, as well as clinical manifestations related to hyperandrogenism. his condition not only leads to reproductive issues but is also linked to psychological disorders, such as depression. The exact etiology of PCOS remains incompletely understood; however, it is suggested that, alongside genetic factors, insulin resistance, an abnormal rise in circulating testosterone levels, and obesity-related inflammation may contribute to ovarian dysfunction.

lifestyle intervention is the current recommendation that could enhance anthropometric indices, cardio-metabolic markers, and reproductive characteristics of women with PCOS. Recent evidence indicated that the administration of lipid-soluble antioxidants may influence lipid profiles and lipid peroxidation levels in individuals with PCOS. Furthermore, previous studies have reported the positive effects of supplementation with antioxidants on other complications associated with PCOS, including inflammatory markers and insulin resistance.

Astaxanthin (ASX) is a carotenoid fat-soluble pigment with potential antioxidant properties naturally found in certain seafood and a specific type of algae. As a consequence of the unique molecular structure of this component, the beneficial effects of ASX on various health aspects involving lipid profile, blood pressure, and depression have been proposed by recent studies . Several experimental investigations also indicated the anti-oxidative and anti-inflammatory impact of ASX supplementation in various PCOS models; however, there are limited studies on the impact of ASX on the cardio-metabolic profile, inflammatory biomarkers, and clinical manifestation of women with PCOS. This paper will describe the design, methodology, and potential clinical implications of the impact of ASX supplementation in women with PCOS.

Thus, this trial aims to investigate the effect of 12 weeks of 10 mg/day astaxanthin administration compared to a control group on insulin sensitivity, lipid profile, circulating Malondialdehyde (MDA) levels, severity of hirsutism, and depression in women with PCOS.

Material and methods Study setting and recruitment This is a single-center double-blind, randomized controlled clinical trial with two parallel groups: one intervention group and one control group. Eligible women with PCOS who are referred to the collaborating gynecologist clinic in Isfahan, Iran, in 2024-2025, will be recruited in this study. After outlining the study's objectives, written informed consent will be obtained from all participants. All participants will be assigned a project-specific code that will be used throughout all data analyses.

Randomization and allocation Data on general information and socio-economic status will be obtained through face-to-face interviews. After recording information at baseline, participants will be randomly divided into two intervention and placebo groups. Using the Permuted Block Randomization method and a table of random numbers, patients will be randomly allocated to receive ASX supplements or placebo after stratifying for age, and metformin intake.

Subjects in the intervention group will receive one capsule containing 10 mg ASX per day made by the "Zyest Technology Tarawat Zendig" institute in Iran. The dosage of ASX is determined based on the safe amount of ASX consumption recorded in the relevant articles. The placebo group will take one capsule containing corn starch in a wrapped and covered form and the appearance of ASX supplementation (blinding). The pharmaceutical company coded both participants in the ASX and placebo groups (codes A and B). The investigators and participants will remain unaware of the allocation, and the code will be kept concealed until the study concludes.

To ensure participant adherence, all women are requested to return the supplement packs at each visit (every two weeks), and the remaining prescribed supplements will be counted within that timeframe. Additionally, the compliance of study participants will be monitored daily through social networks. Participants will be instructed not to alter their common diet and physical activities during the study.

Outcome measures Evaluation of general, demographic, and anthropometric characteristics Participant's general information including age, history of illness, desired disease phenotype (diagnosis by a doctor with the phenotype section in the demographic information questionnaire and smoking will be collected through a general information questionnaire by interview. The questionnaire will be carefully filled with questions from the participant and the patient's contact number will also be recorded. Data collection, including laboratory data, blood pressure, and anthropometric measurements will be assessed at baseline and 12 weeks (post-intervention). For anthropometric evaluations, all measurements will be performed according to the method provided by the World Health Organization. Standing height will be measured using a wall-mounted height meter (Seca 206, Germany) with an accuracy of 0.1 cm without shoes, heels attached to the wall knees straight, looking forward and shoulders in a normal position. A weight measurement of people with minimal clothes and without shoes will be done using a digital scale with an accuracy of 100 grams. BMI will also be calculated by dividing weight (in kilograms) by the square of height (in meters).

Dietary intake assessment The individual's dietary intake will be evaluated using a 24-hour dietary recall in the four scenarios (at the baseline, 4-week, 8-week, and the end of the study) by a trained nutritionist. the reported amounts of each food and drink consumed will be converted to grams per day using the household guidebook. Diet information analysis will be done using Nutritionist IV software (First Databank, Hearst Corp, San Bruno, CA, USA).

Physical Activity Assessment Questionnaire The physical activity evaluation of the participants will be recorded by the short form of the International Physical Activity Questionnaire (IPAQ) 4 times (at the baseline, 4-week, 8-week, and the end of the study). To obtain the overall physical activity score based on MET-minutes/week, the score obtained from 3 activity categories including walking, moderate physical activity, and vigorous physical activity will be recorded.

Blood pressure measurement To measure blood pressure, patients were asked to rest for 10 minutes, then the measurement was done using a mercury sphygmomanometer (Riester, Germany). The blood pressure of each person will be measured twice with a time interval of 10 minutes, in a sitting position, from the right arm and at the level of the heart. The average of these two measurements was considered as the patient's blood pressure. Before taking blood pressure, patients will be asked about smoking or drinking coffee in the previous 2 hours.

Evaluation of the severity of hirsutism To assess the severity of hirsutism, the amount of total body hair in nine sits (upper lip, chin, chest, upper and lower abdomen, thigh, upper and lower back, and upper arm) will be evaluated according to the modified Ferriman-Gallwey (mFG) scoring system. In this system, each body sit will be visually scored on a scale of 0 to 4, and the maximum score of each participant could be 16. The final score of 0 to 3 will be measured as non-hirsutism, 4 to 7 will be considered mild hirsutism, and 8 Up to 11 and 12 to 16 will reflect moderate hirsutism and severe hirsutism, respectively. Subjects will be asked to not use any removing hair methods during the study.

Evaluation of biochemical indicators On days zero (before the start of the intervention) and day 80 (the end of the intervention), 10 cc of blood is taken from the patient in the morning and collected in a plastic tube. It is left with 3,600 revolutions for 3-4 minutes and poured into microtubes containing 0.5 ml. The samples are stored in a freezer at -70°C. To reduce the measurement error, all samplings are done at 8-10 in the morning and in the fasting state. Blood samples taken from patients at the beginning and end of the study are centrifuged for 10 minutes at 300 rpm to separate their serum. Serum values of lipid profile (triglyceride (TG) level, total cholesterol, Low-density lipoprotein cholesterol (LDL-c), and High-density lipoprotein cholesterol (HDL-c) serum) are measured by enzymatic colorimetric method. To measure serum cholesterol, cholesteryl ester enzymes are then added to the solution, and cholesterol oxidase is finally converted into cholesterol-4-en-3-one H₂O₂ and the cholesterol concentration of the sample is obtained using the quinoneimine colorimetric marker. Lipase enzyme is used to measure TG, which converts TG into glycerol and fatty acid. Glycerol turns into glycerol phosphate and finally dihydroxyacetone phosphate, H₂O₂. using the quinoneimine colorimetric indicator, the TG concentration of the sample is obtained. To measure LDL, first, all lipoproteins except Very Low-density lipoprotein cholesterol (VLDL), HDL-c, and chylomicrons are removed, and with the addition of cholesterol esterase, cholesterol oxidase enzymes, H₂O₂ cholestenone is finally made, and LDL-c concentration is obtained by measuring the color resulting from the reaction. To evaluate serum HDL-c, firstly, lipoproteins containing apolipoprotein B such as LDL-c, VLDL, and chylomicron are separated with phosphotungstic acid, magnesium ion, and using quinonimine colorimetric marker and enzyme method, HDL-c concentration of the sample is obtained. Serum glucose is converted to glucuronic acid, H₂O₂ by the activity of glucose oxidase, and the glucose concentration is calculated using the quinonimine indicator. Fasting insulin is measured by the enzyme immunoassay method. Monoclonal antibodies are added to the serum to connect to two epitopes of insulin molecules. After adding buffers, insulin concentration is obtained by measuring light absorption. The HOMA-IR index is used to calculate insulin resistance. To calculate the HOMA-IR index, fasting insulin in the U/mlμ scale and fasting glucose in the /l nmol scale are used: HOMA-IR = fasting insulin (μU/L) x fasting glucose (nmol/L)/22.5. Serum Malondialdehyde (MDA) values are measured by the TBARS method (Arsam Far Biot Company kit) and with a spectrophotometer or fluorimeter.

Masking In this study, the individual conducting the blood test, the one prescribing the supplements, and the person analyzing the data are unaware of the division of participants into two groups: drug and placebo. Since the astaxanthin supplement and placebo are identical in color and shape, patients are also unaware of this division.

Blinding All baseline assessments will be conducted before randomization, and certain assessments will be performed with blinding for group allocation.

Sample size People with polycystic ovary syndrome will be selected by convenience sampling method. The number of samples will be calculated by considering the first type error α=0.05 and the second type error β=0.2 (80% power) and using the following formula.

=((Z_(1-α/2)+Z_(1-β) )^2×〖(S〗_1^2+S_2^2))/d^2 Based on the primary outcome considered on inflammatory factors and by placing the numbers obtained from a study conducted on the effect of astaxanthin supplementation on Malondialdehyde (MDA) [18], the value of d significant difference observed in the level (p < 0.05) and equal to 0.884 mmol/liter will be equal to 17 people in each group, which will be 44 people, including the drop of 25% of people during the study.

Statistical analysis In this study, the quantitative variables will be reported as mean (standard deviation), and qualitative variables will be reported as number (percentage). The evaluation of the normality of the distribution of quantitative variables will be done using the skewness index and the Q-Q plot diagram. Intra-group analyses will be performed using paired t-tests and between-group analyses will be performed using intention-to-treat analysis. The distribution of qualitative variables will be compared between two groups using the chi-square test. SPSS version 22 software will be used to analyze the data with a significance level of P<0.05.

Discussion The complications caused by this disorder are numerous and in addition to clinical symptoms related to hyperandrogenism (such as hirsutism, acne, and androgenic alopecia) and lack of ovulation, metabolic and atherosclerotic complications as well as an increased risk of complications during pregnancy may be observed in these people.

Although, the treatment strategies available for these patients are quite limited, currently, hormonal combination drugs are considered the first line of treatment. However, treatment with hormones may be associated with complications such as increased risk of cardiovascular diseases and high blood pressure. Currently, one of the things that can be useful for patients with PCOS is improving people's lifestyle, including proper dietary interventions and more physical activity, which should be considered in all affected women.

Astaxanthin (ASX) is a carotenoid pigment and a fat-soluble antioxidant found naturally in certain seafood, including shrimp and crab, as well as in specific types of algae. ASX is more active than other carotenoids and, unlike them, converts to vitamin A. due to its unique molecular structure, it has antioxidant properties 500 times stronger than vitamin E. Astaxanthin's ability to regulate immunity and systemic inflammation has been confirmed in many studies. Also, in recent studies, the complementary effects of this antioxidant have been seen to improve blood pressure, lipid profile levels, and systemic inflammation .

Based on a study in 2011 by Choi et al., which was conducted on 27 people with BMI above 25 for 12 weeks, it was found that treatment with astaxanthin decreased LDL-c and Apo B, but no significant changes occurred in other lipid biomarkers. Also, after 12 weeks, the level of MDA and Isoprostan (ISP) decreased in the intervention group, but the total antioxidant capacity (TAC) increased in this group. Therefore, in general, astaxanthin supplementation improved the lipid profile (LDL, Apo B) and oxidative stress. Despite animal studies of the effect of astaxanthin on PCOS, there have been limited human studies in this field. After comparing our study with one of these human studies, it was found that in our study, the patient's lipid profile is one of the important factors and conditions in PCOS patients, blood sugar indicators, which are very important due to the discussion of insulin resistance, and depression index. DASS (the effect that hormonal changes will have on mood) is measured, but none of these factors were measured in the mentioned study. The duration of the study in this article was 60 days, which seemed to be less time compared to the 80 days of our study. Because in such intervention studies, the longer the duration of the intervention, the more valid the results will be. In another study, only TAC (Total antioxidant capacity) level and activation of the Nrf2 axis were measured in PCOS patients. None of the parameters of blood sugar, lipid profile, depression level, and other antioxidant capacities (malondialdehyde) were considered. The duration of the study was 40 days and the dose used was 8 mg. But the length of our study is 80 days and the dose used is 10 mg. Therefore, it will be better and more efficient in terms of value and validity. Our study will not measure indicators such as body mass analysis and other antioxidant capacities. However, this study is one of the first attempts to assess the clinical efficacy of astaxanthin as an auxiliary treatment in PCOS patients. It will provide more evidence in this area.

Declarations Ethics approval and consent to participate The Ethics Committee of Isfahan University of Medical Sciences registered this study. Ethical consent will be obtained from all subjects. This plan is registered on the Iran Clinical Trials (IRCT) website. All participants may withdraw their cooperation from this project at any time, also all participants will be able to request compensation if they suffer harm from the trial. All information obtained from individuals will remain confidential and used only for research purposes, and the patient's identity will remain confidential following the law. All costs related to patient tests, which are outside the periodical tests prescribed by the attending physician, will be borne by the researchers and the organization supporting the project, and the results of the tests will be provided to the individuals at the end of the study. At the end of the study, all the people participating in the research will be thanked in writing. We will publish the results obtained from the study in the form of articles in prestigious international journals.

Consent for publication Not applicable Availability of data and materials The datasets used and/or analyzed during the current study are available from the corresponding author upon reasonable request.

Competing interests The authors declare that they have no competing interests. Funding Isfahan University of Medical Sciences Authors' contributions L.S, N.SH-M, Z.H, S.S Design and analyze data. L.S, M.S, A.A Data collection. M.NJ, N.SH-M major contributor in writing the manuscript. All authors read and approved the final manuscript.

Acknowledgments Not applicable. Patient and Public Involvement Not applicable.

List of abbreviations

PCOS: Polycystic Ovary Syndrome ASX: Astaxanthin MDA: Malondialdehyde IPAQ: International Physical Activity Questionnaire LDL-c: Low-density lipoprotein cholesterol

HDL-c: High-density lipoprotein cholesterol

TG: Triglyceride

VLDL: Very Low-density lipoprotein cholesterol

consent form Study Title: The effectiveness of Astaxanthin supplementation on the clinical symptoms and cardio-metabolic profile in women with Polycystic Ovary Syndrome: A protocol for a randomized double-blinded, placebo-controlled parallel-group study Sponsor's Study ID: Isfahan University of Medical Sciences Study Doctor: Nafiseh Shokri-Mashhadi Email: Nafiseh.shokri@yahoo.com Fax: +9836681378 Postal code: 81746-73461 Sponsor/Funder(s): Isfahan University of Medical Sciences Trial registration number: Iran Clinical Trials (IRCT) website. (IRCT20231001059573N1) Emergency Contact Number (24 hours / 7 days a week): +989171254752 INTRODUCTION You are being invited to participate in a clinical trial (a type of study that involves research). You are invited to participate in this trial because you have Study entry conditions. This consent form provides you with information to help you make an informed choice. Please read this document carefully and ask any questions you may have. All your questions should be answered to your satisfaction before you decide whether to participate in this research study.

Please take your time in making your decision. You may find it helpful to discuss it with your friends and family.

The study staff will tell you about the study timelines for making your decision.

Taking part in this study is voluntary. Deciding not to take part or deciding to leave the study later will not result in any penalty or affect current or future health care.

IS THERE A CONFLICT OF INTEREST? The authors declare that they have no competing interests. WHY IS THIS STUDY BEING DONE? This trial aims to investigate the effect of astaxanthin (ASX) on insulin sensitivity, lipid profile, circulating MDA levels, severity of hirsutism, and depression in women with Polycystic Ovary Syndrome (PCOS).

HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY? It is anticipated that about 44 people will take part in this study, from research sites located in Isfahan, Iran.

This study should take 3 months complete for every participant. WHAT IS THE STUDY INTERVENTION? Evaluation of general, demographic, and anthropometric characteristics Dietary intake assessment Physical Activity Assessment Questionnaire Blood pressure measurement Evaluation of the severity of hirsutism Evaluation of biochemical indicators) Blood sampling (

WHAT ARE THE RESPONSIBILITIES OF STUDY PARTICIPANTS?

If you choose to participate in this study, you will be expected to:

Tell the study doctor about your current medical conditions; Tell the study doctor about all prescription and non-prescription medications and supplements, including vitamins and herbals, and check with the study doctor before starting, stopping or changing any of these. This is for your safety as these may interact with the intervention you receive on this study; Tell the study doctor if you are thinking about participating in another research study; Return any unused study medication; Return any questionnaires that you take home to complete; Tell the study doctor if you become pregnant or father a child while participating on this study; Avoid drinking/eating medicine, supplements ASX supplement is for you alone, and must not be shared with others.

CAN PARTICIPANTS CHOOSE TO LEAVE THE STUDY? You can choose to end your participation in this research (called withdrawal) at any time without having to provide a reason. If you choose to withdraw from the study, you are encouraged to contact the study doctor or study staff.

You may withdraw your permission to use information that was collected about you for this study at any time by letting the study doctor know. However, this would also mean that you withdraw from the study.

CAN PARTICIPATION IN THIS STUDY END EARLY?

The study doctor may stop your participation in the study early, and without your consent, for reasons such as:

The study intervention does not work for you; You are unable to tolerate the study intervention; You are unable to complete all required study procedures; New information shows that the study intervention is no longer in your best interest; The study doctor no longer feels this is the best option for you; The Sponsor decides to stop the study; The Regulatory Authority Research Ethics Board withdraws permission for this study to continue; Your group assignment becomes known to you or others (like the study doctor or study staff); If you plan to, or become, pregnant If this happens, it may mean that you would not receive the study intervention for the full period described in this consent form.

If you are removed from this study, the study doctor will discuss the reasons with you and plans will be made for your continued care outside of the stu

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 45 years
2. Clinical diagnosis of polycystic ovary syndrome
3. Have a body mass index of 25-35 kg/m 2
4. Absence of pregnancy and breastfeeding
5. No intake of medicine
6. Not willing to get pregnant during the study
7. No presence of chronic inflammatory diseases or other endocrine disorders
8. No current treatments except metformin
9. No intake of dietary supplements within at last 2 previous months

Exclusion Criteria:

1. Consuming less than 80% of the total administered ASX supplements
2. Ongoing pregnancy
3. Changing their usual diet or eating habits or level of physical activity
4. Presence of Skin or digestive allergy symptoms or any desired complications by intake of ASX supplementation
5. Smoking or alcohol consumption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — eligible women with PCOS and a body mass index of 25-35 kg/m2, who are referred to the gynecologist clinic in Isfahan, Iran,
Enrollment: 44 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement | From enrollment to the end of treatment at 8 weeks
  To measure blood pressure, patients were asked to rest for 10 minutes, then the measurement was done using a mercury sphygmomanometer (Riester, Germany). The blood pressure of each person will be measured twice with a time interval of 10 minutes, in a sitting position, from the right arm and at the level of the heart. The average of these two measurements was considered as the patient's blood pressure. Before taking blood pressure, patients will be asked about smoking or drinking coffee in the previous 2 hours
Evaluation of the severity of hirsutism | From enrollment to the end of treatment at 8 weeks
  To assess the severity of hirsutism, the amount of total body hair in nine sits (upper lip, chin, chest, upper and lower abdomen, thigh, upper and lower back, and upper arm) will be evaluated according to the modified Ferriman-Gallwey (mFG) scoring system. In this system, each body sit will be visually scored on a scale of 0 to 4, and the maximum score of each participant could be 16. The final score of 0 to 3 will be measured as non-hirsutism, 4 to 7 will be considered mild hirsutism, and 8 Up to 11 and 12 to 16 will reflect moderate hirsutism and severe hirsutism, respectively. Subjects will be asked to not use any removing hair methods during the study.
Evaluation of biochemical indicators | From enrollment to the end of treatment at 8 weeks
  On days zero (before the start of the intervention) and day 80 (the end of the intervention), 10 cc of blood is taken from the patient in the morning and collected in a plastic tube. It is left with 3,600 revolutions for 3-4 minutes and poured into microtubes containing 0.5 ml. The samples are stored in a freezer at -70°C. To reduce the measurement error, all samplings are done at 8-10 in the morning and in the fasting state. Blood samples taken from patients at the beginning and end of the study are centrifuged for 10 minutes at 300 rpm to separate their serum. Serum values of lipid profile (triglyceride (TG) level, total cholesterol, Low-density lipoprotein cholesterol (LDL-c), and High-density lipoprotein cholesterol (HDL-c) serum) are measured by enzymatic colorimetric method. To measure serum cholesterol, cholesteryl ester enzymes are then added to the solution, and cholesterol oxidase is finally converted into cholesterol-4-en-3-one H₂O₂ and the cholesterol concentration of the
Physical Activity Assessment Questionnaire | 4 times (at the baseline, 4-week, 8-week, and the end of the study)
  The physical activity evaluation of the participants will be recorded by the short form of the International Physical Activity Questionnaire (IPAQ) 4 times (at the baseline, 4-week, 8-week, and the end of the study)(22). To obtain the overall physical activity score based on MET-minutes/week, the score obtained from 3 activity categories including walking, moderate physical activity, and vigorous physical activity will be recorded.
Dietary intake assessment | at the baseline, 4-week, 8-week, and the end of the study)
  The individual's dietary intake will be evaluated using a 24-hour dietary recall in the four scenarios (at the baseline, 4-week, 8-week, and the end of the study) by a trained nutritionist. the reported amounts of each food and drink consumed will be converted to grams per day using the household guidebook(20). Diet information analysis will be done using Nutritionist IV software (First Databank, Hearst Corp, San Bruno, CA, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Nafiseh Shokri-Mashhadi, Dr., Study Director — Isfahan University of Medical Sciences
Locations (1):
- Isfahan university of medical sciences, Isfahan, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gharaei R, Alyasin A, Mahdavinezhad F, Samadian E, Ashrafnezhad Z, Amidi F. Randomized controlled trial of astaxanthin impacts on antioxidant status and assisted reproductive technology outcomes in women with polycystic ovarian syndrome. J Assist Reprod Genet. 2022 Apr;39(4):995-1008. doi: 10.1007/s10815-022-02432-0. Epub 2022 Mar 3. PMID 35237893
- [Background] Jabarpour M, Aleyasin A, Nashtaei MS, Lotfi S, Amidi F. Astaxanthin treatment ameliorates ER stress in polycystic ovary syndrome patients: a randomized clinical trial. Sci Rep. 2023 Feb 28;13(1):3376. doi: 10.1038/s41598-023-28956-8. PMID 36854788
- [Background] Choi HD, Kim JH, Chang MJ, Kyu-Youn Y, Shin WG. Effects of astaxanthin on oxidative stress in overweight and obese adults. Phytother Res. 2011 Dec;25(12):1813-8. doi: 10.1002/ptr.3494. Epub 2011 Apr 8. PMID 21480416
- [Background] Papathanasiou G, Georgoudis G, Papandreou M, Spyropoulos P, Georgakopoulos D, Kalfakakou V, Evangelou A. Reliability measures of the short International Physical Activity Questionnaire (IPAQ) in Greek young adults. Hellenic J Cardiol. 2009 Jul-Aug;50(4):283-94. PMID 19622498
- [Background] Brendler T, Williamson EM. Astaxanthin: How much is too much? A safety review. Phytother Res. 2019 Dec;33(12):3090-3111. doi: 10.1002/ptr.6514. Epub 2019 Dec 1. PMID 31788888
- [Background] Kiel IA, Lionett S, Parr EB, Jones H, Roset MAH, Salvesen O, Vanky E, Moholdt T. Improving reproductive function in women with polycystic ovary syndrome with high-intensity interval training (IMPROV-IT): study protocol for a two-centre, three-armed randomised controlled trial. BMJ Open. 2020 Feb 20;10(2):e034733. doi: 10.1136/bmjopen-2019-034733. PMID 32086359
- [Background] Franks S. Controversy in clinical endocrinology: diagnosis of polycystic ovarian syndrome: in defense of the Rotterdam criteria. J Clin Endocrinol Metab. 2006 Mar;91(3):786-9. doi: 10.1210/jc.2005-2501. Epub 2006 Jan 17. PMID 16418209
- [Background] Toktay E, Selli J, Gurbuz MA, Alaca R. Investigation of the effects of astaxanthin in experimental polycystic ovary syndrome (PCOS) in rats. Iran J Basic Med Sci. 2023;26(10):1155-1161. doi: 10.22038/IJBMS.2023.69984.15223. PMID 37736515
- [Background] Mashhadi NS, Zakerkish M, Mohammadiasl J, Zarei M, Mohammadshahi M, Haghighizadeh MH. Astaxanthin improves glucose metabolism and reduces blood pressure in patients with type 2 diabetes mellitus. Asia Pac J Clin Nutr. 2018;27(2):341-346. doi: 10.6133/apjcn.052017.11. PMID 29384321
- [Background] Bjorklund G, Gasmi A, Lenchyk L, Shanaida M, Zafar S, Mujawdiya PK, Lysiuk R, Antonyak H, Noor S, Akram M, Smetanina K, Piscopo S, Upyr T, Peana M. The Role of Astaxanthin as a Nutraceutical in Health and Age-Related Conditions. Molecules. 2022 Oct 23;27(21):7167. doi: 10.3390/molecules27217167. PMID 36363994
- [Background] Tefagh G, Payab M, Qorbani M, Sharifi F, Sharifi Y, Ebrahimnegad Shirvani MS, Pourghazi F, Atlasi R, Shadman Z, Rezaei N, Mohammadi-Vajari E, Larijani B, Ebrahimpur M. Effect of vitamin E supplementation on cardiometabolic risk factors, inflammatory and oxidative markers and hormonal functions in PCOS (polycystic ovary syndrome): a systematic review and meta-analysis. Sci Rep. 2022 Apr 6;12(1):5770. doi: 10.1038/s41598-022-09082-3. PMID 35388031
- [Background] Zhao J, Sui X, Shi Q, Su D, Lin Z. Effects of antioxidant intervention in patients with polycystic ovarian syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Aug 12;101(32):e30006. doi: 10.1097/MD.0000000000030006. PMID 35960093
- [Background] Borzoei A, Rafraf M, Niromanesh S, Farzadi L, Narimani F, Doostan F. Effects of cinnamon supplementation on antioxidant status and serum lipids in women with polycystic ovary syndrome. J Tradit Complement Med. 2017 May 19;8(1):128-133. doi: 10.1016/j.jtcme.2017.04.008. eCollection 2018 Jan. PMID 29322000
- [Background] Badawy A, Elnashar A. Treatment options for polycystic ovary syndrome. Int J Womens Health. 2011 Feb 8;3:25-35. doi: 10.2147/IJWH.S11304. PMID 21339935
- [Background] Panidis D, Tziomalos K, Papadakis E, Katsikis I. Infertility treatment in polycystic ovary syndrome: lifestyle interventions, medications and surgery. Front Horm Res. 2013;40:128-41. doi: 10.1159/000341824. Epub 2012 Oct 18. PMID 24002410
- [Background] Lim SS, Norman RJ, Davies MJ, Moran LJ. The effect of obesity on polycystic ovary syndrome: a systematic review and meta-analysis. Obes Rev. 2013 Feb;14(2):95-109. doi: 10.1111/j.1467-789X.2012.01053.x. Epub 2012 Oct 31. PMID 23114091
- [Background] Sadeeqa S, Mustafa T, Latif S. Polycystic Ovarian Syndrome-Related Depression in Adolescent Girls: A Review. J Pharm Bioallied Sci. 2018 Apr-Jun;10(2):55-59. doi: 10.4103/JPBS.JPBS_1_18. PMID 29962792
- [Background] Diamanti-Kandarakis E, Papavassiliou AG, Kandarakis SA, Chrousos GP. Pathophysiology and types of dyslipidemia in PCOS. Trends Endocrinol Metab. 2007 Sep;18(7):280-5. doi: 10.1016/j.tem.2007.07.004. Epub 2007 Aug 10. PMID 17692530
- [Background] Dubey P, Reddy S, Boyd S, Bracamontes C, Sanchez S, Chattopadhyay M, Dwivedi A. Effect of Nutritional Supplementation on Oxidative Stress and Hormonal and Lipid Profiles in PCOS-Affected Females. Nutrients. 2021 Aug 25;13(9):2938. doi: 10.3390/nu13092938. PMID 34578816
- [Background] Diamanti-Kandarakis E, Kouli CR, Bergiele AT, Filandra FA, Tsianateli TC, Spina GG, Zapanti ED, Bartzis MI. A survey of the polycystic ovary syndrome in the Greek island of Lesbos: hormonal and metabolic profile. J Clin Endocrinol Metab. 1999 Nov;84(11):4006-11. doi: 10.1210/jcem.84.11.6148. PMID 10566641